CLINICAL TRIAL: NCT00787319
Title: Long-Term Non-Interventional Study (NIS) To Investigate The Safety And Effectiveness Of MACUGEN In Patients With Neovascular Age-Related Macular Degeneration Under Conditions Of Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5751032
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Results first posted 2013-08-13 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Age-related Macular Degeneration
Keywords: Ophthalmology; Age-related macular degeneration; outpatients
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AMD
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — Outpatients with age-related macular degeneration (AMD)
  Other Names: observation only

SUMMARY:
To define what procedures were used for the diagnosis and monitoring of the treatment age-related macular degeneration (AMD). What is the effect of the Macugen, compliance with Macugen treatment, safety profile of Macugen, final physician assessment of treatment with Macugen.

DETAILED DESCRIPTION:
no sampling

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old
* patients with neovascular age-related macular degeneration
* enrollment to study is fully on physician decision in compliance with current SPC

Exclusion Criteria:

* Patient who did not meet indication according to SPC Macugen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Czechia (6):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Olomouc
  - Pfizer Investigational Site, Ostrava - Poruba
  - Pfizer Investigational Site, Pilsen
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Ústí nad Labem

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5751032

RESULTS

PARTICIPANT FLOW:
Groups:
- Pegaptanib: Participants with neovascular age-related macular degeneration (AMD) received pegaptanib intravitreal injection in accordance with Summary of Product Characteristics (SmPC) and observed for a period of up to 24 months or early discontinuation.
Period: Overall Study
Arm/Group | Pegaptanib
Started | 108
Completed | 45
Not Completed | 63
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 15
Not completed — Adverse Event | 3
Not completed — Objective progression or relapse | 30
Not completed — Lack of Efficacy | 1
Not completed — Budget exhausted/exceeded | 1
Not completed — Unresponsiveness to visit invitation | 1
Not completed — No health insurance reimbursement | 2
Not completed — Stabilized disease findings | 3
Not completed — Inactive disease | 5

BASELINE CHARACTERISTICS:
Arm/Group | Pegaptanib
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 43

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Visual Acuity (VA) at Final Visit
Description: Visual acuity (VA) measured as viewing distance (distance for participant/distance for normal vision). Viewing distance considered as fraction to calculate decimal VA. Decimal VA data presented as Logarithm of Minimum Angle of Resolution (logMAR), logMAR= -log10 (decimal VA). It measures VA loss; positive values indicated vision loss, while negative values denote normal/better VA and allowed comparison of data using different viewing distances and/or different charts (85 or 100 letters, 85 letter equivalents to decimal VA of 1.0). Results were based on study eye for which medication was given.
Time Frame: Baseline, Final Visit (Week 104 or early termination [ET])
Population: Full analysis set (FAS) included all enrolled participants who received study medication. Missing values were imputed using last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Pegaptanib
Number analyzed (Participants) | 108
logMAR
  Baseline | 0.61 (0.27)
  Change at Final visit | 0.15 (0.37)

2. Secondary Outcome: Change From Baseline in Visual Acuity (VA) at Each Visit
Description: VA measured as viewing distance (distance for participant/distance for normal vision). Viewing distance considered as fraction to calculate decimal VA. Decimal VA data presented as logMAR, logMAR= -log10 (decimal VA). It measures VA loss; positive values indicated vision loss, while negative values denote normal/better VA and allowed comparison of data using different viewing distances and/or different charts (85 or 100 letters, 85 letter equivalents to decimal VA of 1.0). Results were based on study eye for which medication was given.
Time Frame: Baseline, Week 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, 102
Population: FAS included all enrolled participants who received study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies participants evaluated at each time point, respectively.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Pegaptanib
Number analyzed (Participants) | 93
logMAR
  Change at Week 6 (n=93) | -0.03 (0.13)
  Change at Week 12 (n=88) | 0.03 (0.23)
  Change at Week 18 (n=76) | 0.03 (0.27)
  Change at Week 24 (n=75) | 0.01 (0.27)
  Change at Week 30 (n=74) | 0.03 (0.26)
  Change at Week 36 (n=68) | 0.02 (0.29)
  Change at Week 42 (n=59) | 0.06 (0.28)
  Change at Week 48 (n=68) | 0.10 (0.35)
  Change at Week 54 (n=50) | 0.09 (0.35)
  Change at Week 60 (n=46) | 0.10 (0.35)
  Change at Week 66 (n=25) | 0.10 (0.41)
  Change at Week 72 (n=19) | 0.14 (0.51)
  Change at Week 78 (n=20) | 0.19 (0.37)
  Change at Week 84 (n=13) | 0.05 (0.35)
  Change at Week 90 (n=16) | -0.05 (0.24)
  Change at Week 96 (n=11) | -0.10 (0.28)
  Change at Week 102 (n=20) | 0.16 (0.37)

3. Secondary Outcome: Number of Participants With Change in Visual Acuity (VA) as Compared to Previous Examination
Description: VA measured as viewing distance (distance for participant/distance for normal vision). Viewing distance considered as fraction to calculate decimal VA. logMAR= -log10 (decimal VA). It measures VA loss; positive values indicated vision loss,negative values denote normal/better VA and allowed comparison of data using different viewing distances and/or different charts(85 or 100 letters, 85 letter equivalents to decimal VA of 1.0). Results based on study eye for which medication was given. Number of participants with VA improved, unchanged or worsened as compared to previous examination reported.
Time Frame: Week 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, 102
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 90
participants
  Week 6: Improved (n=90) | 20
  Week 6: Unchanged (n=90) | 64
  Week 6: Worsened (n=90) | 6
  Week 12: Improved (n=88) | 12
  Week 12: Unchanged (n=88) | 58
  Week 12: Worsened (n=88) | 18
  Week 18: Improved (n=72) | 12
  Week 18: Unchanged (n=72) | 49
  Week 18: Worsened (n=72) | 11
  Week 24: Improved (n=73) | 16
  Week 24: Unchanged (n=73) | 46
  Week 24: Worsened (n=73) | 11
  Week 30: Improved (n=74) | 9
  Week 30: Unchanged (n=74) | 51
  Week 30: Worsened (n=74) | 14
  Week 36: Improved (n=68) | 11
  Week 36: Unchanged (n=68) | 47
  Week 36: Worsened (n=68) | 10
  Week 42: Improved (n=59) | 8
  Week 42: Unchanged (n=59) | 42
  Week 42: Worsened (n=59) | 9
  Week 48: Improved (n=68) | 12
  Week 48: Unchanged (n=68) | 44
  Week 48: Worsened (n=68) | 12
  Week 54: Improved (n=50) | 8
  Week 54: Unchanged (n=50) | 33
  Week 54: Worsened (n=50) | 9
  Week 60: Improved (n=46) | 1
  Week 60: Unchanged (n=46) | 38
  Week 60: Worsened (n=46) | 7
  Week 66: Improved (n=25) | 3
  Week 66: Unchanged (n=25) | 11
  Week 66: Worsened (n=25) | 11
  Week 72: Improved (n=18) | 4
  Week 72: Unchanged (n=18) | 12
  Week 72: Worsened (n=18) | 2
  Week 78: Improved (n=20) | 2
  Week 78: Unchanged (n=20) | 14
  Week 78: Worsened (n=20) | 4
  Week 84: Improved (n=13) | 2
  Week 84: Unchanged (n=13) | 8
  Week 84: Worsened (n=13) | 3
  Week 90: Improved (n=16) | 4
  Week 90: Unchanged (n=16) | 10
  Week 90: Worsened (n=16) | 2
  Week 96: Improved (n=11) | 5
  Week 96: Unchanged (n=11) | 4
  Week 96: Worsened (n=11) | 2
  Week 102: Improved (n=20) | 3
  Week 102: Unchanged (n=20) | 8
  Week 102: Worsened (n=20) | 9

4. Secondary Outcome: Physician's Assessment of Efficacy
Description: Efficacy was based on the study eye for which pegaptanib treatment was given. Number of participants with each grade of efficacy of treatment, as assessed by the physician was reported on the 5 point categorical scale: excellent, very good, good, fair, poor.
Time Frame: Week 104 or End of study (EOS)
Population: FAS included all enrolled participants who received study medication.
Measure: Number; unit: participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 108
participants
  Excellent | 20
  Very Good | 16
  Good | 24
  Fair | 12
  Poor | 36

5. Other Pre Specified Outcome: Number of Participants With Procedures for Age-related Macular Degeneration (AMD) Diagnosis and Monitoring
Description: Procedures used for diagnosis of AMD and monitoring of the course of treatment included fluorescein angiography (FA), optical coherent tomography (OCT), or other (Ot) procedure apart from FA and OCT. OCT, FA, and other are not mutually exclusive, hence same participant may be included in more than 1 procedure for AMD diagnosis and monitoring at a particular time point.
Time Frame: Baseline, Week 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, 102
Population: Safety analysis set included all enrolled participants who received study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies participants evaluated at each time point, respectively.
Measure: Number; unit: participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 87
participants
  Baseline: Diagnosis,OCT (n=87) | 85
  Baseline: Diagnosis,FA (n=87) | 61
  Baseline: Diagnosis,Ot (n=87) | 12
  Baseline: Monitoring,OCT (n=25) | 25
  Baseline: Monitoring,FA (n=25) | 6
  Baseline: Monitoring,Ot (n=25) | 1
  Week 6: Monitoring,OCT (n=21) | 21
  Week 12: Monitoring,OCT (n=32) | 32
  Week 18: Monitoring,OCT (n=20) | 20
  Week 18: Monitoring,Ot (n=20) | 1
  Week 24: Monitoring,OCT (n=23) | 23
  Week 24: Monitoring,FA (n=23) | 1
  Week 24: Monitoring,Ot (n=23) | 1
  Week 30: Monitoring,OCT (n=20) | 20
  Week 30: Monitoring,Ot (n=20) | 1
  Week 36: Monitoring,OCT (n=21) | 20
  Week 36: Monitoring,Ot (n=21) | 1
  Week 42: Monitoring,OCT (n=14) | 14
  Week 48: Monitoring,OCT (n=19) | 19
  Week 54: Diagnosis,OCT (n=2) | 1
  Week 54: Diagnosis,FA (n=2) | 2
  Week 54: Monitoring,OCT (n=18) | 18
  Week 54: Monitoring,FA (n=18) | 2
  Week 60: Monitoring,OCT (n=13) | 13
  Week 60: Monitoring,FA (n=13) | 1
  Week 60: Monitoring,Ot (n=13) | 1
  Week 66: Monitoring,OCT (n=3) | 3
  Week 72: Monitoring,OCT (n=6) | 6
  Week 72: Monitoring,Ot (n=6) | 1
  Week 78: Monitoring,OCT (n=10) | 10
  Week 78: Monitoring,Ot (n=10) | 2
  Week 84: Monitoring,OCT (n=11) | 10
  Week 84: Monitoring,FA (n=11) | 1
  Week 84: Monitoring,Ot (n=11) | 1
  Week 90: Diagnosis,OCT (n=1) | 1
  Week 90: Diagnosis,Ot (n=1) | 1
  Week 90: Monitoring,OCT (n=10) | 10
  Week 90: Monitoring,Ot (n=10) | 5
  Week 96: Monitoring,OCT (n=8) | 8
  Week 96: Monitoring,Ot (n=8) | 2
  Week 102: Diagnosis,OCT (n=1) | 1
  Week 102: Diagnosis,FA (n=1) | 1
  Week 102: Monitoring,OCT (n=17) | 12
  Week 102: Monitoring,FA (n=17) | 1
  Week 102: Monitoring,Ot (n=17) | 11

6. Other Pre Specified Outcome: Number of Participants Who Discontinued Treatment Due to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Baseline up to Week 104 (EOS)
Population: Safety analysis set included all enrolled participants who received study medication.
Measure: Number; unit: participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 108
participants | 3

7. Other Pre Specified Outcome: Duration of Treatment
Description: Duration of treatment (in weeks) was calculated as: (date of the last injection of study medication minus date of the first injection of study medication plus 1) divided by 7.
Time Frame: Baseline up to Week 104 (EOS)
Population: Safety analysis set included all enrolled participants who received study medication.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Pegaptanib
Number analyzed (Participants) | 108
weeks | 50.33 (29.40)

8. Other Pre Specified Outcome: Mean Number of Doses of Study Medication Received
Time Frame: Baseline up to Week 104 (EOS)
Population: Safety analysis set included all enrolled participants who received study medication.
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Pegaptanib
Number analyzed (Participants) | 108
doses | 7.48 (3.77)

9. Other Pre Specified Outcome: Physician's Assessment of Tolerability
Description: Number of participants with each grade of tolerability of treatment as assessed by physician was evaluated on the five point categorical scale: excellent, very good, good, fair, poor.
Time Frame: Baseline up to Week 104 (EOS)
Population: Safety analysis set included all enrolled participants who received study medication.
Measure: Number; unit: participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 108
participants
  Excellent | 64
  Very Good | 34
  Good | 8
  Fair | 2
  Poor | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pegaptanib
Serious Adverse Events (participants affected / at risk) | 2/108
Other Adverse Events (participants affected / at risk) | 22/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegaptanib (N=108)
Choroidal neovascularisation (Eye disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegaptanib (N=108)
Age-related macular degeneration (Eye disorders) | 4
Choroidal neovascularisation (Eye disorders) | 3
Conjunctivitis (Eye disorders) | 4
Corneal erosion (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Macular oedema (Eye disorders) | 1
Retinal haemorrhage (Eye disorders) | 2
Subretinal fibrosis (Eye disorders) | 1
Drug ineffective (General disorders) | 1
Granuloma (General disorders) | 1
Conjunctivitis bacterial (Infections and infestations) | 1
Keratitis herpetic (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Dizziness (Nervous system disorders) | 1
Therapeutic embolisation (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.